CLINICAL TRIAL: NCT00316199
Title: Phase II Study of Gemcitabine-Paclitaxel 3-Weekly Schedule as First-Line Treatment in Metastatic Breast Cancer After Anthracycline Failure
Brief Title: Efficacy Study of Gemcitabine-Paclitaxel to Treat Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9803; B9E-MC-JHST
Record Dates: First submitted 2006-04-18; First posted 2006-04-20 (Estimated); Results first posted 2009-06-11 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2009-06

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: gemcitabine; Drug: paclitaxel

INTERVENTIONS:
Drug: gemcitabine — 1250 mg/m2, intravenous (IV), day 1 and day 8 every 21 days until disease progression
  Other Names: LY188011; Gemzar
Drug: paclitaxel — 175 mg/m2, intravenous (IV), every 21 days until disease progression

SUMMARY:
The purpose of this study is to determine the response rate to a gemcitabine-paclitaxel combination administered on a 3-weekly schedule in Chinese patients with unresectable, locally recurrent breast cancer or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female patients of Chinese origin with histologically or cytologically proven diagnosis of breast cancer.
* Unresectable, locally recurrent breast cancer or stage IV disease.
* Have at least one measurable lesion as defined by Response Evaluation Criteria In Solid Tumors (RECIST) criteria.
* Performance Status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Scale
* Treatment with an anthracycline-based chemotherapy regimen in the adjuvant/neoadjuvant setting with subsequent disease relapse.

Exclusion Criteria:

* Prior chemotherapy for unresectable, locally advanced breast cancer or metastatic disease.
* Concurrent administration of any other tumor therapy, including cytotoxic chemotherapy, hormonal therapy, and immunotherapy.
* Known or suspected brain metastasis or second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* Active infection or other serious condition.
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-04; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- China (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine + Paclitaxel: Gemcitabine: 1250 mg/m2, intravenous (IV), day 1 and day 8 every 21 days until disease progression.
  Paclitaxel: 175 mg/m2, intravenous (IV), every 21 days until disease progression
Period: Overall Study
Arm/Group | Gemcitabine + Paclitaxel
Started | 60
Completed | 48
Not Completed | 12
Not completed — Adverse Event | 2
Not completed — Death | 8
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine + Paclitaxel
Number analyzed (Participants) | 60
Age Continuous [Mean (Standard Deviation); unit: years] | 46.9 (8.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 0
Region of Enrollment [Number; unit: participants]
  China | 60
Disease Stage at Study Entry [Number; unit: participants] — Stage of disease was determined using American Joint Committee on Cancer Staging Criteria for Breast Cancer. Stages range from Stage 0 to Stage IV. The higher the stage, the more severe the disease.
  participants
    Stage IIIB | 6
    Stage IV | 54
Eastern Cooperative Oncology Group Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  participants
    0 - Fully Active | 30
    1 - Ambulatory, Restricted Strenuous Activity | 30
Menopausal Status [Number; unit: participants]
  Pre-Menopausal | 29
  Peri-Menopausal | 7
  Post Menopausal | 22
  Missing | 2
Pathological Diagnosis [Number; unit: participants]
  Undifferentiated Breast Carcinoma | 1
  Infiltrating Lobular Carcinoma | 0
  Infiltrating Ductal Breast Carcinoma | 55
  Adenocarcinoma | 3
  Comedocarcinoma | 0
  Missing | 1
Race/Ethnicity [Number; unit: participants]
  East Asian (Chinese) | 60
Height [Mean (Standard Deviation); unit: centimeters] | 160.3 (4.35)
Weight [Mean (Standard Deviation); unit: kilograms] | 62.68 (9.518)

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Tumor Response
Description: Best response recorded from the start of treatment until disease progression/recurrence using Response Evaluation Criteria In Solid Tumors (RECIST) criteria that defines when participants improve ("respond"), stay the same ("stable"), or worsen ("progression") during treatment.
Time Frame: baseline to measured progressive disease (tumor assessments were performed every 2 cycles during study therapy, or 3 months during post-therapy until disease progression, or up to 12 months after enrollment)
Population: All enrolled participants diagnosed with metastatic breast cancer, had measurable disease at baseline, and received at least one dose of study drug. Two participants were excluded from analysis because they received chemotherapy for locally advanced/metastatic breast cancer within 6 months prior to enrollment.
Measure: Number; unit: participants
Arm/Group | Gemcitabine + Paclitaxel
Number analyzed (Participants) | 58
participants
  Complete Response (CR) | 2
  Partial Response (PR) | 27
  Stable Disease (SD) | 20
  Progressive Disease (PD) | 7
  Early Death from Malignant Disease | 0
  Death from Toxicity | 0
  Early Death from Other Causes | 0
  Unknown | 2

2. Secondary Outcome: Time to Treatment Failure
Description: Defined as time from enrollment to the date of death due to any cause, measured disease progression, treatment discontinuation for undocumented progression, early treatment discontinuation for toxicity or other reason, or new anticancer treatment started.
Time Frame: baseline to stopping treatment
Population: All enrolled participants. Time to treatment failure for participants who are still participating in the study without treatment failure at the time of analysis will be treated as censored at thte date of the last tumor assessment (3 participants censored).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine + Paclitaxel
Number analyzed (Participants) | 60
months | 4.5 [4.1 to 5.3]

3. Secondary Outcome: Progression-Free Survival
Description: Defined as the time from enrollment to the date of objective disease progression or death on study, whichever occurs first. Censoring was determined based on US-FDA 2005 draft guidance on clinical endpoints.
Time Frame: baseline to measured progressive disease or death (tumor assessments were performed every 2 cycles during study therapy, or 3 months during post-therapy until disease progression, or up to 12 months after enrollment)
Population: All enrolled participants. Forty-two participants were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine + Paclitaxel
Number analyzed (Participants) | 60
months | 7.6 [5.8 to 8.8]

4. Secondary Outcome: Duration of Response
Description: Measured from the time of first documentation of complete response (CR) or partial response (PR), whichever status is first recorded, until the date of objective disease progression or death on study, whichever occurs first, with censoring defined in the same way as for progression-free survival.
Time Frame: time of response to measured progressive disease or death (tumor assessments were performed every 2 cycles during study therapy, or 3 months during post-therapy until disease progression, or up to 12 months after enrollment)
Population: Enrolled participants who were considered responders (had either a complete response or partial response).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine + Paclitaxel
Number analyzed (Participants) | 29
months | 5.6 [4.4 to 7.6]

5. Secondary Outcome: Overall Survival Probability
Description: Original outcome was overall survival = time from date of enrollment to date of death due to any cause. Survival time was censored at date of last contact for participants who were still alive or lost to follow-up. Because only 8 participants had documented death while on study, results are reported as 6- and 12-month overall survival probability.
Time Frame: baseline to date of death from any cause
Population: All enrolled participants. Fifty-two participants were censored.
Measure: Number; unit: percent
Arm/Group | Gemcitabine + Paclitaxel
Number analyzed (Participants) | 60
percent
  6-Month Overall Survival Probability | 97
  12-Month Overall Survival Probability | 87

ADVERSE EVENTS:
Arm/Group | Gemcitabine + Paclitaxel
Serious Adverse Events (participants affected / at risk) | 1
Other Adverse Events (participants affected / at risk) | 59
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Gemcitabine + Paclitaxel
Femur fracture (Injury, poisoning and procedural complications) | 1/60 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Gemcitabine + Paclitaxel
Leukopenia (Blood and lymphatic system disorders) | 42/60 (116)
Neutropenia (Blood and lymphatic system disorders) | 46/60 (115)
Thrombocytopenia (Blood and lymphatic system disorders) | 3/60 (3)
Abdominal pain (Gastrointestinal disorders) | 5/60 (9)
Constipation (Gastrointestinal disorders) | 5/60 (9)
Diarrhoea (Gastrointestinal disorders) | 10/60 (14)
Nausea (Gastrointestinal disorders) | 13/60 (29)
Vomiting (Gastrointestinal disorders) | 13/60 (38)
Fatigue (General disorders) | 19/60 (78)
Pyrexia (General disorders) | 10/60 (13)
Alanine aminotransferase increased (Investigations) | 16/60 (21)
Aspartate aminotransferase increased (Investigations) | 11/60 (15)
Haemoglobin decreased (Investigations) | 4/60 (5)
Neutrophil count decreased (Investigations) | 5/60 (16)
Platelet count decreased (Investigations) | 5/60 (5)
White blood cell count decreased (Investigations) | 6/60 (14)
Anorexia (Metabolism and nutrition disorders) | 9/60 (18)
Hyperglycaemia (Metabolism and nutrition disorders) | 4/60 (4)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3/60 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 21/60 (64)
Myalgia (Musculoskeletal and connective tissue disorders) | 35/60 (82)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5/60 (17)
Headache (Nervous system disorders) | 3/60 (4)
Neuropathy (Nervous system disorders) | 10/60 (11)
Peripheral sensory neuropathy (Nervous system disorders) | 28/60 (74)
Cough (Respiratory, thoracic and mediastinal disorders) | 4/60 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 50/60 (50)
Rash (Skin and subcutaneous tissue disorders) | 10/60 (13)
Flushing (Vascular disorders) | 3/60 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days